CLINICAL TRIAL: NCT02182999
Title: Continuous Wound Infiltration After Hallux Valgus Surgery A Prospective, Randomized, Double-blind and Placebo-controlled Single-center Trial
Brief Title: Continuous Wound Infiltration After Hallux Valgus Surgery
Acronym: CWI-HVS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Rainer Biedermann, MD, MD, PD, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CWI-HVS
Record Dates: First submitted 2014-06-20; First posted 2014-07-08 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2017-11

CONDITIONS: Hallux Valgus
Keywords: Hallux valgus surgery; wound infiltration; pain
MeSH Terms: conditions — Hallux Valgus; Pain | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NaCl 0,9% (Placebo Comparator): Continuous wound infiltration NaCl 0,9% 2 ml/h for first 24 postoperative hours by wound infiltration catheter (InfiltraLong-Katheter 19G x 420mm; Pajunk Medizintechnologie GmbH)
  Interventions: Device: Wound infiltration catheter; Drug: NaCl 0.9%
- Ropivacaine (Active Comparator): Continuous wound infiltration with Ropivacaine 0,2% 2 ml/h for first 24 postoperative hours by wound infiltration catheter (InfiltraLong-Katheter 19G x 420mm; Pajunk Medizintechnologie GmbH)
  Interventions: Device: Wound infiltration catheter; Drug: Ropivacaine 0.2%

INTERVENTIONS:
Device: Wound infiltration catheter — Wound catheter with multiple and laterally aligned holes is inserted through the intact skin via an 16G iv catheter 2 cm proximal-laterally from the proximal end of the dorsomedial skin incision and placed subcutaneously through the wound and medially around the first metatarsal so that the tip projects into the interdigital space 1/2.
  Other Names: InfiltraLong-Katheter 19G x 420mm, Pajunk
Drug: NaCl 0.9% — The catheter is connected to the perfusor line filled with saline 0.9% to allow continuous wound infiltration at a rate of 2 ml/h for 24 hours.
  Other Names: Saline 0.9%
  Arms: NaCl 0,9%
Drug: Ropivacaine 0.2% — The catheter is connected to the perfusor line filled with Ropivacaine 0.2% to allow continuous wound infiltration at a rate of 2 ml/h for 24 hours.
  Other Names: Ropinaest 0.2%
  Arms: Ropivacaine

SUMMARY:
The aim of this study is to investigate the effect of continuous wound infiltration with ropivacaine in comparison to standard pain management after elective distal metatarsal osteotomy for postoperative pain control.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of continuous wound infiltration with ropivacaine in comparison to standard pain management after elective distal metatarsal osteotomy for postoperative pain control. The primary outcome parameters of this study were average pain and peak pain level on the verbal numeric rating scale (NRS; 1-10, higher numbers indicating increasing pain level) during the first 48 hours after surgery. The secondary outcome parameters included postoperative rescue opioid consumption, clinical outcome (AOFAS forefoot score, ROM of MTP joint of the greater toe), incidence of postoperative complications, and patient satisfaction with surgery on a numeric rating scale (1-10).

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a distal metatarsal osteotomy (only Chevron or Scarf) and lateral release of the adductor halluces muscle with/without concomitant osteotomy of the proximal phalanx of the greater toe (Akin) for idiopathic hallux valgus deformity will be included.

Exclusion Criteria:

* hallux valgus surgery other then mentioned above or concomitant other procedures
* denial to participate and give informed consent
* patients with neurological diseases that affect the sensory-motor function
* patients with any short-term (1 month) previous surgery on affected lower extremity
* allergies or other comorbidity that prohibits standardized pain regime (renal insufficiency, severe heart or liver impairment, uncontrolled asthma, history of peptic ulcera )
* patients unwilling to undergo surgery without general anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer G. Biedermann, MD, Principal Investigator — UK für Orthopädie Innsbruck
Locations (1):
- Department of Orthopedic Surgery, Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients undergoing a distal metatarsal osteotomy and lateral release with/without concomitant osteotomy of the proximal phalanx of the greater toe for idiopathic hallux valgus deformity at the Department of Orthopedic Surgery, Medical University of Innsbruck, between May 2014 and March 2017 were screened for eligibility to the study.
Groups:
- NaCl 0,9%: Continuous wound infiltration NaCl 0,9% 2 ml/h for first 24 postoperative hours by wound infiltration catheter (InfiltraLong-Katheter 19G x 420mm; Pajunk Medizintechnologie GmbH)
  InfiltraLong-Katheter 19G x 420mm, Pajunk: Wound catheter with multiple and laterally aligned holes is inserted through the intact skin via an 16G iv catheter 2 cm proximal-laterally from the proximal end of the dorsomedial skin incision and placed subcutaneously through the wound and medially around the first metatarsal so that the tip projects into the interdigital space 1/2.
  NaCl 0,9%: The catheter is connected to the perfusor line filled with saline 0.9% to allow continuous wound infiltration at a rate of 2 ml/h for 24 hours.
- Ropivacaine: Continuous wound infiltration with Ropivacaine 0,2% 2 ml/h for first 24 postoperative hours by wound infiltration catheter (InfiltraLong-Katheter 19G x 420mm; Pajunk Medizintechnologie GmbH)
  InfiltraLong-Katheter 19G x 420mm, Pajunk: Wound catheter with multiple and laterally aligned holes is inserted through the intact skin via an 16G iv catheter 2 cm proximal-laterally from the proximal end of the dorsomedial skin incision and placed subcutaneously through the wound and medially around the first metatarsal so that the tip projects into the interdigital space 1/2.
  Ropivacaine: The catheter is connected to the perfusor line filled with ropivacain 0.2% to allow continuous wound infiltration at a rate of 2 ml/h for 24 hours.
Period: Overall Study
Arm/Group | NaCl 0,9% | Ropivacaine
Started | 25 | 25
Completed | 20 | 22
Not Completed | 5 | 3
Not completed — Adverse Event | 4 | 3
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NaCl 0,9% | Ropivacaine | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (17.2) | 58.0 (13.1) | 55.2 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 25 | 25 | 50
BMI [Mean (Standard Deviation); unit: kg/m²] | 24.0 (4.0) | 25.8 (4.2) | 24.9 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Average Postoperative Numeric Rating Scale (NRS) for Pain
Description: The primary outcome parameters of this study were average pain and peak pain level on the verbal numeric rating scale (NRS; 1-10, higher numbers indicating increasing pain level) during the first 48 hours after surgery. NRS scores for pain were assessed by members of the nursing staff every 4 hours for 48 hours after the procedure (until discharge). Patients were instructed to rate their pain level on a scale from 0 to 10, with 0 meaning "no pain" and 10 indicating "pain as bad as it could be". Average postoperative numeric rating scale (NRS) for pain was calculated for each group (Placebo, Ropivacaine) by adding all postoperative NRS scores of all patients in each group (Placebo, Ropivacaine) to obtain the mean postoperative NRS score.
Time Frame: First 48 postoperative hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NaCl 0,9% | Ropivacaine
Number analyzed (Participants) | 20 | 22
units on a scale | 2.0 (0.7) | 1.9 (0.8)
Statistical Analysis 1: Comparison: NaCl 0,9% vs Ropivacaine; A sample size of 17 patients in each group was previously calculated on the basis of a significance level of .05, a power of 80%, an anticipated pooled standard Deviation (SD) of 1.0 of the mean verbal NRS pain level, and a minimal clinically important difference in the mean verbal NRS pain level of 1.0 points between the groups. Anticipating a loss to follow-up, we planned to recruit a total of 50 patients (25 patients each group); Test type: Superiority; p = 0.596, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.1

2. Primary Outcome: Peak Postoperative Numeric Rating Scale (NRS) for Pain
Description: The primary outcome parameters of this study were average pain and peak pain level on the verbal numeric rating scale (NRS; 1-10, higher numbers indicating increasing pain level) during the first 48 hours after surgery. NRS scores for pain were assessed by members of the nursing staff every 4 hours for 48 hours after the procedure (until discharge). Patients were instructed to rate their pain level on a scale from 0 to 10, with 0 meaning "no pain" and 10 indicating "pain as bad as it could be". Peak postoperative numeric rating scale (NRS) for pain was calculated for each group (Placebo, Ropivacaine) by adding the highest recorded NRS score for pain of all patients in each group (Placebo, Ropivacaine) to obtain the mean peak postoperative NRS score.
Time Frame: First 48 postoperative hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NaCl 0,9% | Ropivacaine
Number analyzed (Participants) | 20 | 22
units on a scale | 3.9 (1.7) | 3.5 (2.0)
Statistical Analysis 1: Comparison: NaCl 0,9% vs Ropivacaine; Test type: Superiority; p = 0.353, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.4

3. Secondary Outcome: American Orthopaedic Foot and Ankle Society Score (AOFAS)
Description: The American Orthopedic Foot and Ankle Society Score (AOFAS-Score, Forefoot Version) is comprised of nine questions and coveres three categories: Pain (40 points), function (50 points) and alignment (10 points). These are all scored together for a total of 100 points. The scale ranges from 0 to 100, with higher values representing a better outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NaCl 0,9% | Ropivacaine
Number analyzed (Participants) | 18 | 21
units on a scale | 75.8 (8.9) | 75.7 (10.8)

4. Secondary Outcome: Patient's Overall Satisfaction With Surgery
Description: Patient satisfaction with surgery was investigated on a numeric rating scale (NRS; scale 0-10) as part of routine examination 6 weeks after the procedure. Higher numbers indicate higher patients satisfaction.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NaCl 0,9% | Ropivacaine
Number analyzed (Participants) | 18 | 21
units on a scale | 9.1 (1.3) | 9.0 (1.3)

5. Secondary Outcome: Patient's Overall Satisfaction With Pain Management
Description: Patient satisfaction with pain management was investigated on a numeric rating scale (NRS; scale 0-10) as part of routine examination 6 weeks after the procedure. Higher numbers indicate higher patients satisfaction.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NaCl 0,9% | Ropivacaine
Number analyzed (Participants) | 18 | 21
units on a scale | 9.3 (1.2) | 9.0 (1.2)

ADVERSE EVENTS:
Time Frame: All patients that participated in the study between May 2014 and April 2017 were monitored and followed for 6 weeks.
Description: Adverse Event Reporting Description does not differ from the clinicaltrials.gov definitions.
Arm/Group | NaCl 0,9% | Ropivacaine
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/25
Other Adverse Events (participants affected / at risk) | 3/25 | 2/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaCl 0,9% (N=25) | Ropivacaine (N=25)
Local dysesthesia (Nervous system disorders) | 0 (0) | 1 (1) — One patient complained about severe diffuse local dysesthesia of the foot, which completely resolved after catheter removal.
Catheter fixed by a suture (Surgical and medical procedures) | 1 (1) | 0 (0) — One revision had to be performed because the wound infiltration catheter was accidentally fixed by a suture.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaCl 0,9% (N=25) | Ropivacaine (N=25)
Catheter dislocation (Surgical and medical procedures) | 3 (3) | 2 (2) — Catheter dislocation occurred in five cases.

LIMITATIONS AND CAVEATS:
Primary outcome parameters were only available for 42 out of 50 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-02-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT02182999/Prot_SAP_000.pdf
  • Informed Consent Form (2014-02-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT02182999/ICF_001.pdf